CLINICAL TRIAL: NCT07014072
Title: Comprehensive Limb Evaluation and Arterial Revascularization With Toe Pressure Optimization Registry
Acronym: CLEAR TOE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2025/006; 2025-A00272-47 (Registry Identifier: Enregistrement RCB - Agence nationale de sécurité du médicament et des produits de santé - FRANCE)
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Critical Limb Ischemia (CLI)
Keywords: CLTI; toe pressure; limb salvage; endovascular revascularization; theatening
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historical cohort (Sham Comparator): 100 patients with CLTI treated in the past 3 years at the same center. Patients in this cohort were treated according to standard clinical practices at the time, without intensive toe pressure evaluation to guide reinterventions, and with reinterventions guided solely by clinical criteria.
  Interventions: Other: data collection
- Prospective cohort (Experimental): 100 patients included prospectively and treated as part of the study. Patients in this cohort will be followed with an intensive toe pressure evaluation approach (TcPO2), guiding reinterventions according to predetermined thresholds (<30 mmHg or decrease >10% from immediate postoperative assessment). This cohort will receive best medical treatment:
  Interventions: Procedure: intensive toe pressure evaluation

INTERVENTIONS:
Procedure: intensive toe pressure evaluation — This measurement is non-invasive, painless and is also carried out as part of the care in the follow-up of critical limb ischemia. It takes place like a blood pressure measurement except that it is carried out at the level of a toe.
  Arms: Prospective cohort
Other: data collection — retrospective data
  Arms: Historical cohort

SUMMARY:
To address the heterogeneity of practices, better understand the outcomes of cricital limb theatening ischemia (CLTI) patients after endovascular interventions, and recognize effective endovascular options for infrapopliteal artery revascularization in CLTI, our prospective registry aims to tackle the critical question of whether intensive toe pressure evaluation, guiding repeat revascularization using predetermined thresholds (<30 mmHg or decrease >10% from immediate postoperative assessment), could optimize outcomes in patients with CLTI.

DETAILED DESCRIPTION:
Cricital limb theatening ischemia (CLTI) represents the most advanced stage of peripheral arterial disease (PAD), leading to high mortality rates and limb loss. A primary endovascular strategy is now preferred for most patients with CLTI who have occlusive disease of the tibial arteries. This is especially true for the elderly, diabetic patients, and those without suitable venous conduits for bypass. Patients with CLTI and infra-popliteal occlusive disease do not always respond well to the provided treatment, but the underlying reasons, particularly in those showing good initial results after endovascular revascularization, remain to be determined.

The literature strongly supports the use of drug-eluting stents (DES) in treating infrapopliteal arteries. DES are associated with significant improvements in patency, reduced rates of restenosis and reintervention, and better Rutherford-Becker classification and healing of trophic disorders. However, contrary to initial expectations, the SAVAL trial, whose data were made public in December 2023, comparing a DES dedicated to infra-popliteal arteries with percutaneous transluminal angioplasty in patients with CLTI, failed to meet its primary efficacy (increased primary patency and reduced major adverse events rate) and safety objectives at 12 months, despite preliminary data suggesting an advantage in using DES for treating short lesions. A possible explanation is the significant heterogeneity of practices, with less than half of the patients receiving optimal medical treatment and intensive follow-up, highlighting the need for a comprehensive review of treatment strategies in this challenging patient population.

The lack of an established objective follow-up protocol for this patient group underscores the need for innovative approaches. Currently, there is no widely available consensus indicator to estimate whether the revascularization provided will be sufficient to prevent amputation. The Delta-Perf study has completed its recruitment and is expected to provide results on foot perfusion analysis in patients with CLTI before and after revascularization and its predictive value on amputation-free survival. However, despite high initial technical success rates for endovascular interventions, early failure of these minimally invasive procedures is common.

Current recommendations support duplex scan monitoring and prophylactic reintervention for asymptomatic graft stenosis to promote long-term patency, but monitoring and reintervention strategies after endovascular management have been left to the practitioner's discretion. There are no ongoing studies to determine if the initial improvement observed in the foot is actually maintained, and there is little evidence to support indications for repeated interventions in CLTI. Clinical follow-up alone may be insufficient to detect restenosis, as patients may remain asymptomatic until the target artery is occluded, similar to venous grafts in bypasses. Likewise, measuring the ankle-brachial index (ABI) alone has limited value, given the difficulty in determining the level of restenosis, technical limitations in diabetic patients with calcified vessels, and variability in correlation with the severity of lesions.

It is likely that there are subgroups of patients who could benefit more than others from early reintervention. Toe pressure, in this context, offers a measurable, non-invasive, and clinically relevant parameter that can be consistently evaluated even in challenging cases, particularly in heavily calcified patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Rutherford category 4 or 5
* Wounds limited to toes or forefoot with a salvageable limb
* Infrapopliteal lesions (infra-popliteal arteries) with >70% stenosis upon visual assessment during initial angiography

Exclusion Criteria:

* Previous or planned major amputation of the target limb
* Untreated aortoiliac/femoropopliteal stenotic disease limiting flow
* History of infrapopliteal bypass on the target limb
* Failure of percutaneous transluminal angioplasty of the target limb (technical failure)
* Absence of angiographic evidence of a patent artery below the ankle ("desert foot")
* Lesions located inside or near an arterial aneurysm
* Life expectancy < 1 year
* Acute limb ischemia
* Septicemia or bacteremia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2027-07-07 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Toe pressure with Systolic pressure measurement device | Day 15, Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  The Systolic pressure measurement device is suitable for the toes, as part of the diagnosis or monitoring of obliterating arteriopathy of the lower limbs, as for the fingers of the hand during assessments relating to arteriovenous fistulas.
  The Systolic pressure measurement device ingeniously uses photoplethysmography (PPG) associated with a unique algorithm developed and patented by Atys Medical. PPG makes it possible to detect, thanks to a photoelectric cell (sensor), variations in blood flow in skin traffic.
  The Systolic pressure measurement deviceputs the measurement of digital pressure pressure within the reach of all the stakeholders concerned (angiologists, nephrologists, diabetologists, vascular surgeons, wound and healing services, etc.).

SECONDARY OUTCOMES:
Evaluation of Survival | Day 15, Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Describe if patient is alive or not
Evaluation of the absence of target lesion occlusion. | Day 15, Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Evaluation of absence of occlusion of the target lesion by Echo-doppler
Evaluation of target lesion revascularization | Day 15, Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Evaluation of target lesion revascularization using Echo doppler
Evaluation of major adverse limb events | Day 15, Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Evaluation of major amputation or major reinterventions including new bypass surgery, bypass revision, or thrombectomy/thrombolysis related to the target lesion
Evaluation ofthe Wound healing with WiFi classification | Day 15, Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  It takes into account the patient's foot wound, ischemia and infection. This system can be used to determine the estimated 1-year risk of amputation and the estimated probability of benefit/need for revascularization. It is a useful, standardized tool that can help determine patient risk and the need for intervention.
Evaluation of the Wound healing with colorimetry scale | Day 15, Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Colorimetry involves analyzing the different colors present in a wound to determine its condition and stage of healing. Each color corresponds to a specific tissue or biological process.

CONTACTS AND LOCATIONS:
Overall Officials: Eric DUCASSE, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Yes
The data is available from Pr DUACSSE. An email can be sent to her so that she can contact the data manager and owner, the Bordeaux University Hospital. The data can be made available after contractual agreement
Supporting Information: Study Protocol, ICF